CLINICAL TRIAL: NCT02250612
Title: A Phase II, Observer Masked, Active Controlled Study of SYL040012 for the Treatment of Elevated Intraocular Pressure in Patients With Open-angle Glaucoma or Ocular Hypertension
Brief Title: SYL040012, Treatment for Open Angle Glaucoma
Acronym: SYLTAG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sylentis, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYL040012_IV; 2013-002947-27 (EudraCT Number)
Record Dates: First submitted 2014-09-05; First posted 2014-09-26 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: SYL040012; bamosiran; siRNA; RNAi; Glaucoma; Ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- SYL040012 (bamosiran) 0.375% eye drops (Experimental): 1 drop in each eye once daily for 28 consecutive days
  Interventions: Drug: 1 drop of 0.375% SYL040012 (bamosiran)
- SYL040012 (bamosiran) 0.750% eye drops (Experimental): 1 drop in each eye once daily for 28 consecutive days
  Interventions: Drug: 1 drop of 0.750% SYL040012 (bamosiran)
- SYL040012 (bamosiran) 1.125% eye drops (Experimental): 1 drop in each eye once daily for 28 consecutive days
  Interventions: Drug: 1 drop of 1.125% SYL040012 (bamosiran)
- SYL040012 (bamosiran) 1.5% eye drops (Experimental): 1 drop in each eye once daily for 28 consecutive days
  Interventions: Drug: 1 drop of 1.5% SYL040012 (bamosiran)
- Timolol maleate 0.5% ophthalmic solution (Active Comparator): 1 drop in each eye twice daily for 28 consecutive days
  Interventions: Drug: 1 drop of 0.5 % timolol maleate

INTERVENTIONS:
Drug: 1 drop of 0.375% SYL040012 (bamosiran)
  Arms: SYL040012 (bamosiran) 0.375% eye drops
Drug: 1 drop of 0.750% SYL040012 (bamosiran)
  Arms: SYL040012 (bamosiran) 0.750% eye drops
Drug: 1 drop of 1.125% SYL040012 (bamosiran)
  Arms: SYL040012 (bamosiran) 1.125% eye drops
Drug: 1 drop of 1.5% SYL040012 (bamosiran)
  Arms: SYL040012 (bamosiran) 1.5% eye drops
Drug: 1 drop of 0.5 % timolol maleate
  Arms: Timolol maleate 0.5% ophthalmic solution

SUMMARY:
The purpose of this double-masked, randomized, controlled study is to assess the safety and ocular hypotensive efficacy of four different doses of SYL040012 (bamosiran) eye drops compared to Timolol maleate 0.5% after 28 treatment days in patients with elevated intraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of either sex
* Good or fair general health as assessed by the investigator.
* Signed informed consent prior to any clinical trial-related procedures
* Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT)
* Post-washout mean IOP above target range
* BCVA 1.0 logMAR or better by ETDRS in each eye (equivalent to 20/200)
* Stable visual field
* Central corneal thickness 480-620 μm
* Shaffer gonioscopic grade of ≥ 3 (in at least 3 quadrants) in both eyes

Exclusion Criteria:

* Pregnant or breastfeeding females
* Females of childbearing potential not willing to use a medically acceptable contraceptive method
* Clinically significant systemic disease
* Changes of systemic medication that could have a substantial effect on IOP
* Known hypersensitivity to any component of the formulations
* Unable to comply with the clinical trial requirements
* Clinically significant abnormalities in laboratory tests
* Severe visual field defect
* Any secondary glaucoma
* Pseudoexfoliation or pigment dispersion component, history of angle closure or narrow angles.
* IOP ≥ 35 mm Hg in any eye
* Previous non-laser glaucoma surgery or glaucoma laser procedures (e.g., laser trabeculoplasty) and refractive surgery
* Any ocular surgery or laser treatment, cataract extraction or ocular trauma within 6 months prior to Baseline
* Evidence of ocular infection, inflammation, clinically significant blepharitis or conjunctivitis at baseline (Visit 0), or a history of herpes simplex keratitis
* Clinically significant ocular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (4):
  - Sall Research Medical Center, Artesia, California
  - North Bay Eye Associates, Petaluma, California
  - Eye Care Centers Management, Inc (Clayton Eye Center), Morrow, Georgia
  - Taustin Eye Center, Louisville, Kentucky
- Estonia (3):
  - East Tallin Central Hospital, Tallinn
  - Eye Clinic Dr. Krista Turman, Tallinn
  - Tartu University Hospital, Tartu
- Germany (5):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - University Clinic Magdeburg, Magdeburg
  - Klinikum der Universität München, München
  - Universitätsklinikum Münster, Münster
  - University Hospital Regensburg, Regensburg
- Spain (9):
  - Hospital de Torrevieja, Torrevieja, Alicante
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Hospital Clinic, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Instituto de Oftalmobiología Aplicada, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza

RESULTS

PARTICIPANT FLOW:
Groups:
- SYL040012 (Bamosiran) 0.375% Eye Drops: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) 0.375 %
- SYL040012 (Bamosiran) 0.750 % Eye Drops: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) 0.750 %
- SYL040012 (Bamosiran) 1.125% Eye Drops: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) 1.125%
- SYL040012 (Bamosiran) 1.5% Eye Drops: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) 1.5%
- Timolol Maleate 0.5% Ophthalmic Solution: 1 drop in each eye twice daily for 28 consecutive days
  1 drop of timolol maleate: 0.5 %
Period: Overall Study
Arm/Group | SYL040012 (Bamosiran) 0.375% Eye Drops | SYL040012 (Bamosiran) 0.750 % Eye Drops | SYL040012 (Bamosiran) 1.125% Eye Drops | SYL040012 (Bamosiran) 1.5% Eye Drops | Timolol Maleate 0.5% Ophthalmic Solution
Started | 37 | 40 | 37 | 33 | 37
Completed | 36 | 38 | 35 | 33 | 36
Not Completed | 1 | 2 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SYL040012 (Bamosiran) Eye Drops Dose A: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) Dose A
- SYL040012 (Bamosiran) Eye Drops Dose B: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) Dose B
- SYL040012 (Bamosiran) Eye Drops Dose C: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) Dose C
- SYL040012 (Bamosiran) Eye Drops Dose D: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) Dose D
- Total: Total of all reporting groups
Arm/Group | SYL040012 (Bamosiran) Eye Drops Dose A | SYL040012 (Bamosiran) Eye Drops Dose B | SYL040012 (Bamosiran) Eye Drops Dose C | SYL040012 (Bamosiran) Eye Drops Dose D | Timolol Maleate 0.5% Ophthalmic Solution | Total
Number analyzed (Participants) | 37 | 40 | 37 | 33 | 37 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.4) | 59.4 (12.9) | 61.5 (10.1) | 62.4 (11.1) | 60.2 (11.5) | 60.8 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 22 | 24 | 24 | 119
  Male | 12 | 16 | 15 | 9 | 13 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean Diurnal IOP Within Each Treatment Arm
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- SYL040012 (Bamosiran) 0.375 % Eye Drops: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) 0.375 %
- SYL040012 (Bamosiran) 0.75 % Eye Drops: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) 0.75%
Arm/Group | SYL040012 (Bamosiran) 0.375 % Eye Drops | SYL040012 (Bamosiran) 0.75 % Eye Drops | SYL040012 (Bamosiran) 1.125% Eye Drops | SYL040012 (Bamosiran) 1.5% Eye Drops | Timolol Maleate 0.5% Ophthalmic Solution
Number analyzed (Participants) | 36 | 38 | 35 | 33 | 35
mmHg | -2.4 (2.6) | -3.2 (3.9) | -3.1 (2.5) | -3.1 (3.2) | -6.1 (2.2)
Statistical Analysis 1: Comparison: SYL040012 (Bamosiran) 1.125% Eye Drops vs SYL040012 (Bamosiran) 1.5% Eye Drops; Test type: Superiority; p = 0.93, ANCOVA
Statistical Analysis 2: Comparison: SYL040012 (Bamosiran) 0.75 % Eye Drops vs SYL040012 (Bamosiran) 1.5% Eye Drops; Test type: Superiority; p = 0.92, ANCOVA
Statistical Analysis 3: Comparison: SYL040012 (Bamosiran) 0.375 % Eye Drops vs SYL040012 (Bamosiran) 1.5% Eye Drops; Test type: Superiority; p = 0.23, ANCOVA
Statistical Analysis 4: Comparison: SYL040012 (Bamosiran) 0.75 % Eye Drops vs SYL040012 (Bamosiran) 1.125% Eye Drops; Test type: Superiority; p = 0.85, ANCOVA
Statistical Analysis 5: Comparison: SYL040012 (Bamosiran) 0.375 % Eye Drops vs SYL040012 (Bamosiran) 1.125% Eye Drops; Test type: Superiority; p = 0.25, ANCOVA
Statistical Analysis 6: Comparison: SYL040012 (Bamosiran) 0.375 % Eye Drops vs SYL040012 (Bamosiran) 0.75 % Eye Drops; Test type: Superiority; p = 0.18, ANCOVA

2. Secondary Outcome: Change From Baseline in the Mean Diurnal IOP Within Each Treatment Arm
Time Frame: Baseline and Day 14
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- SYL040012 (Bamosiran) Eye Drops 1.125%: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) 1.125%
- SYL040012 (Bamosiran) Eye Drops 0.75%: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) 0.75%
Arm/Group | SYL040012 (Bamosiran) 1.5% Eye Drops | SYL040012 (Bamosiran) Eye Drops 1.125% | SYL040012 (Bamosiran) Eye Drops 0.75% | SYL040012 (Bamosiran) 0.375 % Eye Drops | Timolol Maleate 0.5% Ophthalmic Solution
Number analyzed (Participants) | 36 | 38 | 35 | 33 | 35
mmHg | -2.4 (2.6) | -2.9 (2.4) | -2.5 (2.1) | -2.4 (3.1) | -5.8 (1.9)
Statistical Analysis 1: Comparison: SYL040012 (Bamosiran) 1.5% Eye Drops vs SYL040012 (Bamosiran) Eye Drops 1.125%; Test type: Superiority; p = 0.94, ANCOVA
Statistical Analysis 2: Comparison: SYL040012 (Bamosiran) 1.5% Eye Drops vs SYL040012 (Bamosiran) Eye Drops 0.75%; Test type: Superiority; p = 0.38, ANCOVA
Statistical Analysis 3: Comparison: SYL040012 (Bamosiran) 1.5% Eye Drops vs SYL040012 (Bamosiran) 0.375 % Eye Drops; Test type: Superiority; p = 0.85, ANCOVA
Statistical Analysis 4: Comparison: SYL040012 (Bamosiran) Eye Drops 1.125% vs SYL040012 (Bamosiran) Eye Drops 0.75%; Test type: Superiority; p = 0.412, ANCOVA
Statistical Analysis 5: Comparison: SYL040012 (Bamosiran) Eye Drops 1.125% vs SYL040012 (Bamosiran) 0.375 % Eye Drops; Test type: Superiority; p = 0.79, ANCOVA
Statistical Analysis 6: Comparison: SYL040012 (Bamosiran) Eye Drops 0.75% vs SYL040012 (Bamosiran) 0.375 % Eye Drops; Test type: Superiority; p = 0.28, ANCOVA

3. Secondary Outcome: Change From Baseline in the Glaucoma Quality of Life Questionnaire (GQL-15) Scores Within Each Treatment Arm
Description: The GQL-15 is a 15 item, 4-domain tool. GQL-15 scoring ranges from 0 to 75. Higher scores indicate poorer quality of life.
Time Frame: Baseline and Day 29
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- SYL040012 (Bamosiran) 0.75% Eye Drops: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) 0.75%
- SYL040012 (Bamosiran) Eye Drops 0.375%: 1 drop in each eye once daily for 28 consecutive days
  1 drop of SYL040012 (bamosiran) 0.375%
Arm/Group | SYL040012 (Bamosiran) 1.5% Eye Drops | SYL040012 (Bamosiran) 1.125% Eye Drops | SYL040012 (Bamosiran) 0.75% Eye Drops | SYL040012 (Bamosiran) Eye Drops 0.375% | Timolol Maleate 0.5% Ophthalmic Solution
Number analyzed (Participants) | 36 | 38 | 35 | 33 | 35
units on a scale | 20 (8.28) | 20.7 (7.68) | 19.4 (6.34) | 22 (9.65) | 18.7 (6.21)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | SYL040012 (Bamosiran) Eye Drops Dose A | SYL040012 (Bamosiran) Eye Drops Dose B | SYL040012 (Bamosiran) Eye Drops Dose C | SYL040012 (Bamosiran) Eye Drops Dose D | Timolol Maleate 0.5% Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/40 | 0/37 | 0/33 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/40 | 0/37 | 0/33 | 0/37
Other Adverse Events (participants affected / at risk) | 4/37 | 9/40 | 6/37 | 2/33 | 2/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYL040012 (Bamosiran) Eye Drops Dose A (N=37) | SYL040012 (Bamosiran) Eye Drops Dose B (N=40) | SYL040012 (Bamosiran) Eye Drops Dose C (N=37) | SYL040012 (Bamosiran) Eye Drops Dose D (N=33) | Timolol Maleate 0.5% Ophthalmic Solution (N=37)
Headache (Nervous system disorders) | 1 (1) | 1 (5) | 3 (3) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (2) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Eye pruritus (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Instillation site pain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No